CLINICAL TRIAL: NCT05800392
Title: A National, Single Center, Randomized, Prospective, Phase IV, Double-blind, Placebo-controlled, Parallel Study to Assess the Efficacy and Safety of DEC103 in the Pain Control Associated With Intrauterine Device (IUD) Insertion
Brief Title: Efficacy and Safety of DEC103 in Pain Control Associated to Intrauterine Device (IUD) Insertion
Acronym: DEC103
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEC103-IV-0123
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain
Keywords: Pain; IUD insertion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): DEC103: The participants will take 02 (two) pills of the sublingual formulation and 01 (one) pill of the oral one, 1 hour prior the IUD insertion.
  Interventions: Drug: DEC103
- Placebo (Placebo Comparator): PLACEBO DEC103: The participants will take 02 (two) pills of the placebo sublingual formulation and 01 (one) pill of the placebo oral one, 1 hour prior the IUD insertion.
  Interventions: Drug: Placebo DEC103

INTERVENTIONS:
Drug: DEC103 — The intervention is composed by two medications: An active sublingual pill and an active oral one.
  Arms: Experimental
Drug: Placebo DEC103 — The intervention is composed by two medications: A placebo sublingual pill and an placebo oral one.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DEC103 in the pain control associated with IUD insertion in women with 18 to 49 years.

DETAILED DESCRIPTION:
The DEC103 treatment is composed by two different medications that are already available in brazilian market. One is a sublingual pill and the other is an oral one. The participants must take 02 (two) pills of the sublingual formulation and 01 (one) of the oral formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent to participate in the study prior to admission;
* Female patients aged between 18 and 49 years old;
* First IUD users;
* Nulliparous women.

Exclusion Criteria:

* Any finding or clinical observation (clinical/physical evaluation) or laboratory condition that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical trial or presence of uncontrolled chronic disease(s);
* Presence of chronic pelvic pain and any uterine malformation;
* Presence of psychiatric disorder;
* Chronic use of medications that interfere with the pain threshold, for example: antidepressants and anticonvulsants;
* Use of analgesics and/or ant-inflammatory in the last 24 hours prior the procedure;
* Any sign or symptom of vaginal or cervical infection;
* Participants with any contraindication to one or both medicines that constitute the DEC103 treatment;
* Actual abuse of alcohol or drugs;
* Participants who are nursing;
* Presence of known allergy or hypersensitivity to the components of the drugs used during the clinical trial;
* Participants with a current medical history of cancer and/or cancer treatment in the last five (05) years;
* Participation in a clinical research protocol in the last 12 months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator judges that there may be a direct benefit to it.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of DEC103 in pain management associated to IUD insertion assessed by NRS. | During the procedure.
  Mean pain during the IUD insertion procedure during IUD deployment. The pain will be assessed through a Numeric Rating Scale (NRS), numbered from 0 (no pain) to 10 (worst pain possible).
Efficacy of DEC103 in pain management associated to IUD insertion assessed by NRS. | During the procedure.
  Mean overall pain rating during the IUD insertion procedure. The pain will be assessed through a Numeric Rating Scale (NRS), numbered from 0 (no pain) to 10 (worst pain possible).
Efficacy of DEC103 in pain management associated to IUD insertion assessed by NRS. | 10 minutes after de procedure.
  Mean pain 10 minuts after the IUD insertion The pain will be assessed through a Numeric Rating Scale (NRS), numbered from 0 (no pain) to 10 (worst pain possible).

SECONDARY OUTCOMES:
Efficacy of DEC103 in pain associated to IUD insertion assessed by NRS. | During the procedure.
  Mean pain during tenaculum placement and uterine sounding. The pain will be assessed through a Numeric Rating Scale (NRS), numbered from 0 (no pain) to 10 (worst pain possible).
Women's overall pain perception during the procedure assessed by a 4-point scale. | During the procedure.
  The global pain perception during the procedure will be assessed through a 4-point scale as the following: 0 = no pain; 1 = mild pain; 2 = moderate pain; 3 = intense pain
Physician's perception regarding ease of IUD insertion assessed by the following options: easy, moderate and difficult. | Immediately after the procedure.
  Physician's perception will be assessed through a questionnaire with the following options: easy, moderate and difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Bahamondes, MD, Principal Investigator — Center for Research on Reproductive Health of Campinas
Locations (1):
- CEMICAMP - Centro de Pesquisas em Saúde Reprodutiva de Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No